CLINICAL TRIAL: NCT03166280
Title: Evaluation of Vitamin D and Iron Status in Chronic Hepatitis C Virus Patients Before and After Treatment
Brief Title: Hepatitis c and Vitamin D and Iron Status
Acronym: hepatitisc
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Eman Sayed Hassan Abd Allah (Other)
Responsible Party: Sponsor-Investigator, Eman Sayed Hassan Abd Allah, principle investigator, assistant professor of Medical Physiology, Assiut University
Organization: Assiut University (Other)
Other Study IDs: IRB0000871820032017
Record Dates: First submitted 2017-05-14; First posted 2017-05-25 (Actual); Last update posted 2017-05-25 (Actual); Status verified 2017-05

CONDITIONS: Hepatitis C
Keywords: hepatitis C; vitamin D; iron; hepcidin
MeSH Terms: conditions — Hepatitis C | interventions — Sofosbuvir; daclatasvir

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- hepatitisC-pre-ttt: Naïve HCV Patients (>18Y) coming to National Committee for control of viral hepatitis before receiving their treatment
- hepatitis C-ttt: Naïve HCV Patients (>18Y) coming to National Committee for control of viral hepatitis- 12 weeks after stoppage their treatment of sofosbuvir 400 mg/day plus Daclatasvir 60 mg/day for 12 weeks.
  Interventions: Drug: Sofosbuvir 400 mg; Drug: Daclatasvir 60 mg/day

INTERVENTIONS:
Drug: Sofosbuvir 400 mg — treatment for hepatitis c by sofosbuvir (Sovaldi) 400 mg/day
  Other Names: sovaldi
  Groups: hepatitis C-ttt
Drug: Daclatasvir 60 mg/day — treatment for hepatitis c by Daclatasvir 60 mg/day
  Other Names: Daklinza
  Groups: hepatitis C-ttt

SUMMARY:
HCV is associated with vitamin D deficiency. Iron overload is frequently occurred in chronic hepatitis C patients; more than one third of HCV positive patients have elevated serum iron, ferritin, and transferrin which were linked to bad prognosis. Hepcidin is a regulatory peptide that is mainly synthesized by the liver cells and plays an important role in iron homeostasis. There is an interaction between iron metabolism and vitamin D metabolism. Iron is essential for vitamin D activation and vitamin D deficiency is associated with elevated hepcidin level, which partly accounts for anemia associated with vitamin D deficiency. Up to our knowledge, little is known about the association between vitamin D status and iron metabolism in HCV patients.

DETAILED DESCRIPTION:
Hepatitis C virus (HCV) is one of the global public health problems. World Health Organization (WHO) reported that more than 80 million people all over the world are infected with HCV. Approximately 700000 persons die every year from hepatitis C-related complications. Egypt is one of the highest prevalence rates of HCV, worldwide.

Vitamin D possesses anti-inflammatory, anti-oxidant, anti-fibrotic and immunomodulatory effects. HCV is associated with vitamin D deficiency. Liver plays an important role in vitamin D hydroxylation and iron metabolism. It stores iron, synthesizes iron transporting protein (transferrin), iron storage protein (ferritin) and an iron regulatory peptide (hepcidin). Iron overload is frequently occurred in chronic hepatitis C patients. More than one third of HCV positive patients have elevated serum iron, ferritin, and transferrin which were linked to bad prognosis. Excess iron is catalyzed by the rapid Fenton reaction producing hydroxyl radicals from hydrogen peroxide and superoxide (10), which induces lipid peroxidation and cellular damage. Hepcidin is a regulatory peptide that is mainly synthesized by the liver cells and plays an important role in iron homeostasis via inhibiting iron absorption and preventing iron efflux from macrophages and thus prevents normal recycling of the iron needed for erythropoiesis. In addition, hepcidin inhibits HCV replication via activation of STAT3. A reduced serum hepcidin has been reported in chronic HCV patients which was correlated to the severity of liver histopathological changes and related to iron overload in these patients.

There is an interaction between iron metabolism and vitamin D metabolism. Iron is essential for vitamin D activation and vitamin D deficiency is associated with elevated hepcidin level, which partly accounts for anemia associated with vitamin D deficiency. Up to our knowledge, little is known about the association between vitamin D status and iron metabolism in HCV patients.

ELIGIBILITY:
Inclusion Criteria:

• Naïve HCV Patients (>18Y) coming to National Committee for control of viral hepatitis to receive their treatment

Exclusion Criteria:

* Age less than 18 years old or more than 70 years old.
* previously received treatment for HCV
* Manifestations or history of manifestations of liver cell failure and cirrhosis including ascites and hepatic encephalopathy.
* Patients co-infected by the hepatitis B (HBV), human immunodeficiency viruses (HIV).
* Hepatocellular carcinoma and other extra hepatic carcinoma.
* Renal disease.
* Patients receiving vitamin D, calcium therapy or iron supplementation for the last 3 months will be excluded.
* Total serum bilirubin ≥ 3 mg/dl.
* Serum albumin < 2.8 g/dl
* international normalization ratio (INR)> 1.7
* Platelet count <50000/mm3
* Serum creatinine >2.5mg/l

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hepatitis C ttt sofobuvir & daclatasvir
Sampling Method: Non-Probability Sample
Enrollment: 87 (Estimated)
Dates: Start 2017-06 (Estimated); Primary Completion 2017-11 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
change in levels of vitamin D | 6 months
  Serum vitamin D (25OH vitamin D) before starting the treatment and after 6 months
Change in iron level | 6 months
  Serum iron level before treatment and after 6 months
Change in total iron binding capacity | 6 month
  Serum total iron binding capacity before starting the treatment and after 6 months
Change in serum hepcidin | 6 months
  Serum hepcidin before starting the treatment and after 6 months

SECONDARY OUTCOMES:
correlate levels of vitamin D, iron, total iron binding capacity and hepcidin with sustain virologic response or any complications | one day
  pearson's correlation

CONTACTS AND LOCATIONS:
Overall Officials: Eman SH Abd Allah, PHD, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided